CLINICAL TRIAL: NCT00650767
Title: A Study of ARRY-438162 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARRAY-162-201
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ARRY-438162 (Schedule 1) (Experimental)
  Interventions: Drug: ARRY-438162, MEK inhibitor; oral
- ARRY-438162 (Schedule 2) (Experimental)
  Interventions: Drug: ARRY-438162, MEK inhibitor; oral
- ARRY-438162 (Schedule 3) (Experimental)
  Interventions: Drug: ARRY-438162, MEK inhibitor; oral
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; oral

INTERVENTIONS:
Drug: ARRY-438162, MEK inhibitor; oral — multiple dose, single schedule
  Arms: ARRY-438162 (Schedule 1); ARRY-438162 (Schedule 2); ARRY-438162 (Schedule 3)
Drug: Placebo; oral — matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2 study, involving a 12-week treatment period, designed to evaluate the effectiveness of investigational study drug ARRY-438162 in treating rheumatoid arthritis in patients on stable doses of methotrexate, and to further evaluate the safety of the study drug. Approximately 200 patients from the US, Argentina, Brazil, Hungary, Peru, Poland and Romania will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of rheumatoid arthritis, based on the American College of Rheumatology (ACR) 1987 Revised Criteria, prior to first dose of study drug.
* Patient has received a stable dose of methotrexate for ≥ 6 weeks prior to first dose of study drug and is willing to continue on this regimen for the duration of the study.
* Patient has received a stable dose of folate for ≥ 6 weeks and is willing to continue on this regimen for the duration of the study.
* No prior use of biological agents for the treatment of rheumatoid arthritis.
* Additional criteria exist.

Key Exclusion Criteria:

* Diagnosis of any other inflammatory or non-inflammatory arthritis that may interfere with disease activity assessments or clinically apparent osteoarthritis which would affect subsequent efficacy measures.
* A history of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological disease or severe systemic involvement with rheumatoid arthritis.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- Spartanburg Medical Research, Spartanburg, South Carolina, United States
- Argentina (6):
  - Asistencia Integral en Reumatologia, Buenos Aires
  - CEMIC, Buenos Aires
  - Hospital Britanico, Buenos Aires
  - CER San Juan, San Juan
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán
  - Centro de Investigaciones Clinicas del Litoral SRL, Santa Fe
- Brazil (7):
  - Médicos Unidos Ltda., Goiânia, Goiás
  - CETI - Hospital das Clínicas da Universidade Federal do Paraná, Curitiba, Paraná
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da da Pontifícia Universidade Católica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital São Paulo / Instituto Paulista de Reumatologia, São Paulo, São Paulo
  - Hospital Heliópolis, São Paulo, São Paulo
  - Instituto de Medicina Avançada (IMA Brasil), São Paulo, São Paulo
- Hungary (7):
  - Budai Irgalmasrendi Kórház - Allergólógia és Immunológia, Budapest
  - Synexus Ltd Hungary, Budapest
  - Békés Megyei Pándy Kálmán Kórház - Rheumatology, Gyula
  - Mozgasszervi Rehabilitacios Kozpont, Mezőkövesd
  - Fejér Megyei Szent György Kórház - Rheumatology, Székesfehérvár
  - MÁV Kórház - Clinical Pharmacology, Szolnok
  - Vas Megyei Markusovszky Korhaz Lajos Általános, Rehabilitációs és Gyógyfürdő Kórház, Egyetemi Oktató Kórház, Zártkörűen Működő Nonprofit Részvénytársaság - Rheumatology, Szombathely
- Peru (4):
  - Instituto de Investigacion y Seguridad Medica EIRL, Arequipa
  - Clinica San Felipe - Centro de Estudios Clinicos CGYM, Lima
  - Clínica Ricardo Palma- Sitio de Investigacion de Reumatologia, Lima
  - Hospital Maria Auxiliadora - Centro de Investigaciones Medicas, Lima
- Poland (6):
  - Centrum Osteoporozy i Chorób Kostno-Stawowych, Bialystok
  - Wojewódzki Szpital Zespolony - Oddział Reumatologiczny, Elblag
  - Centrum Leczenia Chorob Cywilizacyjnych, Gdynia
  - NZOZ Reumed, Lublin
  - Centrum Leczenia Chorob Cywilizacyjnych, Warsaw
  - Synexus SCM Sp. z o.o., Wroclaw
- Romania (4):
  - Spitalul Clinic "Sf, Maria", Bucharest
  - Spitalul Clinic Judetean de Urgenta, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta, Târgu Mureş
  - Cabinet Medical "Prof. Dr. Miorara Banciu", Timișoara

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The ARRAY-162-201 study began recruitment on 04-April-2008 (First Patient First Visit) and concluded on 07-July-2009 (Last Patient Last Visit).
  This study was conducted at 36 sites in the United States, Europe and South America.
Pre-assignment Details: Participant Flow and Baseline Demographics represent the Intent-to-Treat (ITT) population, which is all patients who were randomized to a treatment group.
Groups:
- Placebo: Placebo tablets were identical in appearance to both the 10 mg and 20 mg ARRY-438162 tablets.
  Patients were randomized in a 1:1:1:1 fashion to ARRY-438162 10 mg bid, 40 mg qd or 20 mg bid, or placebo.
- ARRY-438162: 10 mg Bid; ARRY-438162: 40 mg qd; ARRY-438162: 20 mg Bid: Patients were randomized in a 1:1:1:1 fashion to ARRY-438162 10 mg bid, 40 mg qd or 20 mg bid, or placebo.
Period: Overall Study
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Started | 51 | 50 | 50 | 50
Completed | 46 | 41 | 36 | 39
Not Completed | 5 | 9 | 14 | 11
Not completed — Adverse Event | 0 | 3 | 10 | 8
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 3 | 3
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Other | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Demographics represent the Intent-to-Treat (ITT) population, which is all patients who were randomized to a treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid | Total
Number analyzed (Participants) | 51 | 50 | 50 | 50 | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 43 | 45 | 41 | 45 | 174
  >=65 years | 8 | 5 | 9 | 5 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (12.67) | 51.6 (11.98) | 54.8 (11.88) | 51.4 (11.74) | 52.6 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 42 | 43 | 44 | 172
  Male | 8 | 8 | 7 | 6 | 29
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic Or Latino | 24 | 21 | 23 | 24 | 92
  Not Hispanic Or Latino | 27 | 29 | 27 | 26 | 109
Weight [Mean (Standard Deviation); unit: kilogram] | 74.1 (18.26) | 68.2 (14.17) | 72.1 (17.95) | 67.2 (13.86) | 69.2 (15.49)
Height [Mean (Standard Deviation); unit: centimeters] | 160.2 (8.63) | 159.5 (8.11) | 158.6 (9.22) | 158.0 (7.44) | 158.7 (8.25)
Smoking Status [Number; unit: participants]
  Current Smoker | 6 | 10 | 9 | 12 | 37
  Never Smoked | 38 | 39 | 36 | 36 | 149
  Past Smoker | 7 | 1 | 5 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology 20% (ACR20) Response Rate at Week 12
Description: The ACR (American College of Rheumatology) Criteria is a standard criteria to measure the effectiveness of various arthritis medications or treatments in clinical trials for Rheumatoid Arthritis.
  The ACR 20 has a positive outcome if 20% improvement in tender or swollen joint counts were achieved as well as a 20% improvement in at least three of the other five criteria.
Time Frame: Week 12
Population: Analysis group is comprised of the Intent-to-Treat (ITT) population, which is all patients who were randomized to a treatment group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 51 | 50 | 50 | 50
percentage of participants | 45.1 [31.1 to 59.7] | 58.0 [43.2 to 71.8] | 60.0 [45.2 to 73.6] | 54.0 [39.3 to 68.2]

2. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response Rate at Week 1
Description: as for outcome 1
Time Frame: Week 1
Population: Analysis group is comprised of the Efficacy Evaluable population, which is all randomized patients who had at least one post-Baseline assessment of at least one efficacy endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 12.2 [4.6 to 24.8] | 20.8 [10.5 to 35.0] | 32.7 [19.9 to 47.5] | 46.0 [31.8 to 60.7]

3. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response Rate at Week 2
Description: as for outcome 1
Time Frame: Week 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 18.4 [8.8 to 32.0] | 31.3 [18.7 to 46.3] | 32.7 [19.9 to 47.5] | 50.0 [35.5 to 64.5]

4. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response Rate at Week 4
Description: as for outcome 1
Time Frame: Week 4
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 44.9 [30.7 to 59.8] | 54.2 [39.2 to 68.6] | 44.9 [30.7 to 59.8] | 58.0 [43.2 to 71.8]

5. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response Rate at Week 8
Description: as for outcome 1
Time Frame: Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 49.0 [34.4 to 63.7] | 56.3 [41.2 to 70.5] | 53.1 [38.3 to 67.5] | 48.0 [33.7 to 62.6]

6. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response Rate at Week 16 (Follow-up)
Description: as for outcome 1
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 40.8 [27.0 to 55.8] | 52.1 [37.2 to 66.7] | 49.0 [34.4 to 63.7] | 46.0 [31.8 to 60.7]

7. Secondary Outcome: American College of Rheumatology 50% (ACR50) Response Rate at Week 1
Description: The ACR (American College of Rheumatology) Criteria is a standard criteria to measure the effectiveness of various arthritis medications or treatments in clinical trials for Rheumatoid Arthritis.
  The ACR 50 has a positive outcome if 50% improvement in tender or swollen joint counts were achieved as well as a 50% improvement in at least three of the other five criteria.
Time Frame: Week 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 2.0 [0.1 to 10.9] | 6.3 [1.3 to 17.2] | 2.0 [0.1 to 10.9] | 4.0 [0.5 to 13.7]

8. Secondary Outcome: American College of Rheumatology 50% (ACR50) Response Rate at Week 2
Description: as for outcome 7
Time Frame: Week 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 6.1 [1.3 to 16.9] | 8.3 [2.3 to 20.0] | 10.2 [3.4 to 22.2] | 16.0 [7.2 to 29.1]

9. Secondary Outcome: American College of Rheumatology 50% (ACR50) Response Rate at Week 4
Description: as for outcome 7
Time Frame: Week 4
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 10.2 [3.4 to 22.2] | 8.3 [2.3 to 20.0] | 12.2 [4.6 to 24.8] | 16.0 [7.2 to 29.1]

10. Secondary Outcome: American College of Rheumatology 50% (ACR50) Response Rate at Week 8
Description: as for outcome 7
Time Frame: Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 16.3 [7.3 to 29.7] | 27.1 [15.3 to 41.8] | 16.3 [7.3 to 29.7] | 22.0 [11.5 to 36.0]

11. Secondary Outcome: American College of Rheumatology 50% (ACR50) Response Rate at Week 12
Description: as for outcome 7
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 24.5 [13.3 to 38.9] | 25.0 [13.6 to 39.6] | 22.4 [11.8 to 36.6] | 22.0 [11.5 to 36.0]

12. Secondary Outcome: American College of Rheumatology 50% (ACR50) Response Rate at Week 16 (Follow-up)
Description: as for outcome 7
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 16.3 [7.3 to 29.7] | 27.1 [15.3 to 41.8] | 30.6 [18.3 to 45.4] | 14.0 [5.8 to 26.7]

13. Secondary Outcome: American College of Rheumatology 70% (ACR70) Response Rate at Week 1
Description: The ACR (American College of Rheumatology) Criteria is a standard criteria to measure the effectiveness of various arthritis medications or treatments in clinical trials for Rheumatoid Arthritis.
  The ACR 70 has a positive outcome if 70% improvement in tender or swollen joint counts were achieved as well as a 70% improvement in at least three of the other five criteria.
Time Frame: Week 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 0.0 [0.0 to 7.3] | 2.1 [0.1 to 11.1] | 0.0 [0.0 to 7.3] | 2.0 [0.1 to 10.6]

14. Secondary Outcome: American College of Rheumatology 70% (ACR70) Response Rate at Week 2
Description: as for outcome 13
Time Frame: Week 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 2.0 [0.1 to 10.9] | 4.2 [0.5 to 14.3] | 0.0 [0.0 to 7.3] | 2.0 [0.1 to 10.6]

15. Secondary Outcome: American College of Rheumatology 70% (ACR70) Response Rate at Week 4
Description: as for outcome 13
Time Frame: Week 4
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 0.0 [0.0 to 7.3] | 4.2 [0.5 to 14.3] | 2.0 [0.1 to 10.9] | 2.0 [0.1 to 10.6]

16. Secondary Outcome: American College of Rheumatology 70% (ACR70) Response Rate at Week 8
Description: as for outcome 13
Time Frame: Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 4.1 [0.5 to 14.0] | 4.2 [0.5 to 14.3] | 4.1 [0.5 to 14.0] | 4.0 [0.5 to 13.7]

17. Secondary Outcome: American College of Rheumatology 70% (ACR70) Response Rate at Week 12
Description: as for outcome 13
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 8.2 [2.3 to 19.6] | 12.5 [4.7 to 25.2] | 8.2 [2.3 to 19.6] | 6.0 [1.3 to 16.5]

18. Secondary Outcome: American College of Rheumatology 70% (ACR70) Response Rate at Week 16 (Follow-up)
Description: as for outcome 13
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
percentage of participants | 6.1 [1.3 to 16.9] | 6.3 [1.3 to 17.2] | 6.1 [1.3 to 16.9] | 10.0 [3.3 to 21.8]

19. Secondary Outcome: American College of Rheumatology (ACR) Response Criteria - Tender Joint Count (28)
Description: The ACR (American College of Rheumatology) Criteria is a standard criteria to measure the effectiveness of various arthritis medications or treatments in clinical trials for Rheumatoid Arthritis.
  Tender joint count is calculated based on the tenderness response of 28 joints. Possible values ranged from 0 to 28. A lower score indicated less joint tenderness.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 16.8 (6.44) | 14.8 (5.49) | 15.0 (5.98) | 17.0 (5.95)

20. Secondary Outcome: American College of Rheumatology (ACR) Response Criteria - Tender Joint Count (28)
Description: as for outcome 19
Time Frame: Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 14.9 (6.81) | 11.6 (6.24) | 11.6 (6.46) | 11.1 (5.84)

21. Secondary Outcome: American College of Rheumatology (ACR) Response Criteria - Tender Joint Count (28)
Description: as for outcome 19
Time Frame: Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 12.3 (6.50) | 10.2 (6.49) | 11.4 (6.31) | 10.0 (6.00)

22. Secondary Outcome: American College of Rheumatology (ACR) Response Criteria - Tender Joint Count (28)
Description: as for outcome 19
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 11.6 (7.46) | 9.0 (6.31) | 9.6 (6.84) | 8.9 (6.02)

23. Secondary Outcome: American College of Rheumatology (ACR) Response Criteria - Tender Joint Count (28)
Description: as for outcome 19
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 9.9 (7.21) | 8.1 (7.04) | 8.3 (6.27) | 7.5 (5.50)

24. Secondary Outcome: American College of Rheumatology (ACR) Response Criteria - Tender Joint Count (28)
Description: as for outcome 19
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 9.4 (7.09) | 7.1 (7.05) | 7.8 (7.50) | 7.8 (6.57)

25. Secondary Outcome: American College of Rheumatology (ACR) Response Criteria - Tender Joint Count (28)
Description: as for outcome 19
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 9.1 (7.13) | 7.4 (7.15) | 9.2 (7.37) | 8.9 (6.97)

26. Secondary Outcome: American College of Rheumatology (ACR) Response Criteria - Swollen Joint Count (28)
Description: The ACR (American College of Rheumatology) Criteria is a standard criteria to measure the effectiveness of various arthritis medications or treatments in clinical trials for Rheumatoid Arthritis.
  The swollen joint count was calculated based on the swelling response of 28 joints. Possible values ranged from 0 to 28. A lower score indicated less joint swelling.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 12.7 (4.45) | 11.4 (4.10) | 12.3 (4.96) | 13.0 (5.31)

27. Secondary Outcome: American College of Rheumatology (ACR) Response Criteria - Swollen Joint Count (28)
Description: as for outcome 26
Time Frame: Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 11.3 (5.72) | 8.0 (4.65) | 9.6 (4.80) | 9.1 (4.96)

28. Secondary Outcome: American College of Rheumatology (ACR) Response Criteria - Swollen Joint Count (28)
Description: as for outcome 26
Time Frame: Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 9.4 (5.45) | 6.9 (4.98) | 8.7 (4.58) | 7.3 (5.76)

29. Secondary Outcome: American College of Rheumatology (ACR) Response Criteria - Swollen Joint Count (28)
Description: as for outcome 26
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 7.9 (5.14) | 5.8 (4.00) | 7.0 (4.70) | 7.1 (6.03)

30. Secondary Outcome: American College of Rheumatology (ACR) Response Criteria - Swollen Joint Count (28)
Description: as for outcome 26
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 6.7 (5.25) | 5.5 (4.64) | 6.9 (5.51) | 6.5 (5.96)

31. Secondary Outcome: American College of Rheumatology (ACR) Response Criteria - Swollen Joint Count (28)
Description: as for outcome 26
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 6.3 (5.67) | 5.3 (4.86) | 6.3 (5.54) | 6.3 (5.92)

32. Secondary Outcome: American College of Rheumatology (ACR) Response Criteria - Swollen Joint Count (28)
Description: as for outcome 26
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 6.5 (5.69) | 4.8 (4.63) | 6.9 (5.72) | 6.5 (5.96)

33. Secondary Outcome: Patient's Assessment of Arthritis Pain - Visual Analog Scale (VAS)
Description: The Patient's Assessment of Pain utilized a 0 to 100 mm visual analog scale, 0 being no pain and 100 being most severe pain.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 68.7 (18.94) | 61.9 (20.32) | 62.4 (21.42) | 63.0 (18.95)

34. Secondary Outcome: Patient's Assessment of Arthritis Pain - Visual Analog Scale (VAS)
Description: as for outcome 33
Time Frame: Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 61.5 (25.16) | 47.9 (22.94) | 48.4 (22.53) | 42.6 (20.62)

35. Secondary Outcome: Patient's Assessment of Arthritis Pain - Visual Analog Scale (VAS)
Description: as for outcome 33
Time Frame: Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 56.5 (23.89) | 46.4 (22.61) | 47.7 (25.20) | 39.6 (22.60)

36. Secondary Outcome: Patient's Assessment of Arthritis Pain - Visual Analog Scale (VAS)
Description: as for outcome 33
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 50.3 (23.78) | 44.5 (25.23) | 44.8 (24.48) | 39.0 (19.75)

37. Secondary Outcome: Patient's Assessment of Arthritis Pain - Visual Analog Scale (VAS)
Description: as for outcome 33
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 49.7 (26.53) | 46.1 (24.97) | 46.4 (25.42) | 41.5 (23.39)

38. Secondary Outcome: Patient's Assessment of Arthritis Pain - Visual Analog Scale (VAS)
Description: as for outcome 33
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 45.9 (28.15) | 43.9 (27.39) | 43.8 (26.93) | 42.3 (21.46)

39. Secondary Outcome: Patient's Assessment of Arthritis Pain - Visual Analog Scale (VAS)
Description: as for outcome 33
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 50.7 (27.93) | 47.1 (26.32) | 48.7 (27.09) | 48.5 (23.93)

40. Secondary Outcome: Patient's Global Assessment of Arthritis - Visual Analog Score (VAS)
Description: The Patient's Global Assessment of Arthritis was an evaluation based on the patient's disease signs, functional capacity and physical examination, and was independent of the Physician's Global Assessment of Arthritis. The patient self-assessed how the arthritis affected their lives at the time of the visit using the visual analog scale (VAS).
  Patients answered the following: "Considering all the ways in which illness and health conditions may affect you at this time, please make a mark below to show how you are doing." The patient's response was recorded using the 100 mm visual analog scale between 0 (Very Well) and 100 (Very Poorly).
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 65.2 (20.59) | 60.1 (20.80) | 63.4 (19.25) | 55.4 (20.34)

41. Secondary Outcome: Patient's Global Assessment of Arthritis - Visual Analog Score (VAS)
Description: as for outcome 40
Time Frame: Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 57.2 (24.52) | 45.8 (22.65) | 48.3 (22.82) | 42.3 (20.66)

42. Secondary Outcome: Patient's Global Assessment of Arthritis - Visual Analog Score (VAS)
Description: as for outcome 40
Time Frame: Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 57.6 (21.74) | 46.3 (23.62) | 49.4 (22.61) | 40.3 (22.33)

43. Secondary Outcome: Patient's Global Assessment of Arthritis - Visual Analog Score (VAS)
Description: as for outcome 40
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 50.5 (23.96) | 43.5 (24.57) | 46.7 (23.70) | 40.0 (20.55)

44. Secondary Outcome: Patient's Global Assessment of Arthritis - Visual Analog Score (VAS)
Description: as for outcome 40
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 48.7 (26.34) | 42.9 (24.69) | 45.5 (22.95) | 41.8 (21.60)

45. Secondary Outcome: Patient's Global Assessment of Arthritis - Visual Analog Score (VAS)
Description: as for outcome 40
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 45.5 (26.71) | 40.6 (23.24) | 43.4 (24.82) | 41.1 (19.75)

46. Secondary Outcome: Patient's Global Assessment of Arthritis - Visual Analog Score (VAS)
Description: as for outcome 40
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 46.9 (26.69) | 42.6 (22.99) | 47.5 (27.18) | 44.8 (21.95)

47. Secondary Outcome: Physician's Global Assessment of Arthritis - Visual Analog Score (VAS)
Description: The Physician's Global Assessment of Arthritis was an evaluation based on the patient's disease signs, functional capacity and physical examination, and was independent of the Patient's Global Assessment of Arthritis. The Investigator assessed how the overall arthritis appeared at the time of the visit using the visual analog scale (VAS).
  The physician's response was recorded using the 100 mm visual analog scale between 0 (Very Good) and 100 (Very Bad).
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 61.2 (16.71) | 66.0 (13.80) | 61.0 (15.23) | 59.7 (13.26)

48. Secondary Outcome: Physician's Global Assessment of Arthritis - Visual Analog Score (VAS)
Description: as for outcome 47
Time Frame: Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 53.7 (17.80) | 47.7 (19.55) | 46.8 (18.21) | 41.1 (17.14)

49. Secondary Outcome: Physician's Global Assessment of Arthritis - Visual Analog Score (VAS)
Description: as for outcome 47
Time Frame: Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 47.9 (18.61) | 41.8 (18.67) | 43.9 (19.45) | 35.3 (18.27)

50. Secondary Outcome: Physician's Global Assessment of Arthritis - Visual Analog Score (VAS)
Description: as for outcome 47
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 42.0 (19.83) | 39.9 (21.55) | 38.8 (18.40) | 34.7 (19.20)

51. Secondary Outcome: Physician's Global Assessment of Arthritis - Visual Analog Score (VAS)
Description: as for outcome 47
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 39.5 (20.96) | 37.0 (21.21) | 36.8 (18.88) | 32.7 (22.50)

52. Secondary Outcome: Physician's Global Assessment of Arthritis - Visual Analog Score (VAS)
Description: as for outcome 47
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 35.8 (21.96) | 34.9 (22.19) | 35.7 (21.06) | 31.2 (21.64)

53. Secondary Outcome: Physician's Global Assessment of Arthritis - Visual Analog Score (VAS)
Description: as for outcome 47
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 36.7 (20.86) | 33.2 (19.22) | 40.7 (21.92) | 34.6 (20.37)

54. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI)
Description: The HAQ-DI contains a list of items that assessed the degree of difficulty experienced in 8 categories of daily living activities (included in 20 questions) over the past week: Dressing and grooming, arising, eating, walking, hygiene, reach, grip and other activities. Each activity category consists of 2 or 3 items. For each question in the HAQ-DI, the level of difficulty was scored from 0 to 3 with 0 equal to "without difficulty," 1 equal to "with some difficulty," 2 equal to "with much difficulty" and 3 equal to "unable to do." Any activity that required assistance from another individual or required the use of an assistive device adjusted to a minimum score of 2 to represent a more limited functional status.
  The HAQ-DI score takes values between 0 and 3, with a higher score indicating greater disability.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 1.6 (0.59) | 1.5 (0.52) | 1.5 (0.53) | 1.5 (0.65)

55. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI)
Description: as for outcome 54
Time Frame: Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 1.6 (0.66) | 1.3 (0.58) | 1.3 (0.63) | 1.2 (0.68)

56. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI)
Description: as for outcome 54
Time Frame: Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 1.5 (0.59) | 1.3 (0.59) | 1.3 (0.62) | 1.0 (0.62)

57. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI)
Description: as for outcome 54
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 1.4 (0.63) | 1.3 (0.68) | 1.2 (0.63) | 1.1 (0.60)

58. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI)
Description: as for outcome 54
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 1.4 (0.70) | 1.2 (0.72) | 1.2 (0.62) | 1.1 (0.66)

59. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI)
Description: as for outcome 54
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 1.3 (0.72) | 1.1 (0.66) | 1.1 (0.68) | 1.1 (0.64)

60. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI)
Description: as for outcome 54
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 1.3 (0.76) | 1.2 (0.70) | 1.2 (0.64) | 1.1 (0.62)

61. Secondary Outcome: C-Reactive Protein (CRP) at Baseline
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
mg/dL | 1.9 (1.42) | 1.8 (1.18) | 2.4 (1.86) | 2.4 (1.95)

62. Secondary Outcome: C-Reactive Protein (CRP) at Week 1
Time Frame: Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
mg/dL | 2.2 (2.20) | 1.9 (2.85) | 2.0 (2.17) | 1.4 (1.58)

63. Secondary Outcome: C-Reactive Protein (CRP) at Week 2
Time Frame: Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
mg/dL | 1.9 (1.70) | 1.9 (1.70) | 2.5 (2.36) | 2.1 (2.07)

64. Secondary Outcome: C-Reactive Protein (CRP) at Week 4
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
mg/dL | 1.9 (1.55) | 2.2 (3.18) | 2.6 (3.02) | 2.2 (2.25)

65. Secondary Outcome: C-Reactive Protein (CRP) at Week 8
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
mg/dL | 2.1 (2.24) | 2.0 (1.88) | 2.6 (2.39) | 3.0 (3.34)

66. Secondary Outcome: C-Reactive Protein (CRP) at Week 12
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
mg/dL | 2.1 (2.14) | 1.8 (1.87) | 2.5 (2.51) | 2.9 (2.91)

67. Secondary Outcome: C-Reactive Protein (CRP) at Week 16 (Follow-up)
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
mg/dL | 1.9 (1.79) | 2.3 (3.33) | 2.0 (1.68) | 2.3 (2.50)

68. Secondary Outcome: Disease Activity Score (DAS) Using C-Reactive Protein (DAS28-4[CRP])
Description: The DAS28-4(CRP) score is a measure of the subject's disease activity. DAS28-4(CRP) is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity and CRP. DAS28 provides a number on a scale (0 to 10) indicating current disease activity. A score above 5.1 means high disease activity and a score below 3.2 indicates low disease activity.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 6.1 (0.77) | 5.9 (0.61) | 6.0 (0.79) | 6.1 (0.77)

69. Secondary Outcome: Disease Activity Score (DAS) Using C-Reactive Protein (DAS28-4[CRP])
Description: as for outcome 68
Time Frame: Week 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 5.8 (1.01) | 5.0 (1.03) | 5.2 (1.08) | 5.0 (0.97)

70. Secondary Outcome: Disease Activity Score (DAS) Using C-Reactive Protein (DAS28-4[CRP])
Description: as for outcome 68
Time Frame: Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 5.4 (0.94) | 4.9 (1.17) | 5.3 (1.06) | 4.8 (1.14)

71. Secondary Outcome: Disease Activity Score (DAS) Using C-Reactive Protein (DAS28-4[CRP])
Description: as for outcome 68
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 5.2 (1.13) | 4.7 (1.28) | 5.0 (1.19) | 4.7 (1.24)

72. Secondary Outcome: Disease Activity Score (DAS) Using C-Reactive Protein (DAS28-4[CRP])
Description: as for outcome 68
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 4.9 (1.23) | 4.6 (1.34) | 4.8 (1.15) | 4.6 (1.40)

73. Secondary Outcome: Disease Activity Score (DAS) Using C-Reactive Protein (DAS28-4[CRP])
Description: as for outcome 68
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 4.8 (1.26) | 4.3 (1.39) | 4.6 (1.42) | 4.6 (1.43)

74. Secondary Outcome: Disease Activity Score (DAS) Using C-Reactive Protein (DAS28-4[CRP])
Description: as for outcome 68
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 4.8 (1.20) | 4.4 (1.27) | 4.8 (1.42) | 4.7 (1.42)

75. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Physical Functioning
Description: The SF-36v2 (Acute version) is a 36-item generic health status measure that yields an 8-scale profile of functional health and well-being as well as psychometrically-based physical and mental health summary measures.
  The SF-36v2 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. The lower the score the more disability, while the higher the score the less disability.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 29.8 (8.45) | 31.4 (7.78) | 31.6 (8.29) | 33.8 (9.58)

76. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Physical Functioning
Description: as for outcome 75
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 33.8 (9.05) | 36.0 (9.10) | 34.3 (9.73) | 38.7 (8.74)

77. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Physical Functioning
Description: as for outcome 75
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 34.2 (9.86) | 37.2 (9.25) | 34.9 (10.32) | 38.2 (10.36)

78. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Physical Functioning
Description: as for outcome 75
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 34.5 (11.08) | 37.2 (9.83) | 36.4 (10.91) | 38.8 (9.63)

79. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Physical Functioning
Description: as for outcome 75
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 35.4 (11.10) | 36.0 (9.75) | 35.5 (8.99) | 37.8 (9.84)

80. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Role-Physical
Description: as for outcome 75
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 30.3 (8.47) | 32.7 (8.07) | 32.3 (7.68) | 32.9 (8.49)

81. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Role-Physical
Description: as for outcome 75
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 34.8 (8.20) | 37.1 (9.69) | 37.1 (7.89) | 38.6 (7.88)

82. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Role-Physical
Description: as for outcome 75
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 34.6 (9.17) | 39.2 (9.70) | 36.5 (8.09) | 39.2 (9.20)

83. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Role-Physical
Description: as for outcome 75
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 35.1 (9.65) | 39.7 (10.36) | 37.9 (9.46) | 39.3 (8.12)

84. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Role-Physical
Description: as for outcome 75
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 36.4 (10.45) | 38.9 (8.50) | 36.9 (9.48) | 38.7 (9.21)

85. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Bodily Pain
Description: as for outcome 75
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 32.5 (6.39) | 33.1 (6.22) | 32.4 (7.18) | 33.0 (6.50)

86. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Bodily Pain
Description: as for outcome 75
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 37.3 (8.49) | 38.1 (9.22) | 38.0 (8.58) | 41.0 (9.22)

87. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Bodily Pain
Description: as for outcome 75
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 37.2 (9.05) | 39.1 (9.73) | 38.7 (8.27) | 40.8 (10.11)

88. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Bodily Pain
Description: as for outcome 75
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 38.1 (10.01) | 39.3 (9.21) | 38.7 (9.61) | 40.9 (9.62)

89. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Bodily Pain
Description: as for outcome 75
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 37.9 (10.62) | 38.1 (9.89) | 37.0 (9.73) | 38.1 (9.19)

90. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - General Health
Description: as for outcome 75
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 34.1 (6.65) | 33.6 (8.05) | 34.0 (7.85) | 36.1 (7.44)

91. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - General Health
Description: as for outcome 75
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 36.4 (6.00) | 36.9 (9.10) | 36.9 (9.11) | 38.9 (9.07)

92. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - General Health
Description: as for outcome 75
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 36.8 (7.96) | 37.8 (9.10) | 36.9 (8.21) | 39.7 (9.29)

93. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - General Health
Description: as for outcome 75
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 37.8 (6.93) | 37.1 (9.13) | 36.7 (9.28) | 39.2 (8.74)

94. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - General Health
Description: as for outcome 75
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 37.4 (8.60) | 36.8 (9.02) | 36.4 (8.53) | 38.3 (9.25)

95. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Vitality
Description: as for outcome 75
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 40.1 (10.10) | 41.5 (7.79) | 41.3 (9.17) | 44.5 (8.30)

96. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Vitality
Description: as for outcome 75
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 44.3 (8.75) | 46.3 (10.31) | 44.7 (9.16) | 47.3 (9.64)

97. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Vitality
Description: as for outcome 75
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 43.9 (9.76) | 47.2 (11.08) | 45.3 (10.03) | 49.0 (9.30)

98. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Vitality
Description: as for outcome 75
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 45.5 (9.73) | 47.8 (10.20) | 46.3 (10.56) | 47.5 (9.41)

99. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Vitality
Description: as for outcome 75
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 45.1 (10.55) | 47.4 (11.67) | 44.4 (9.91) | 46.9 (9.93)

100. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Social Functioning
Description: as for outcome 75
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 32.7 (10.97) | 34.1 (9.28) | 34.7 (9.50) | 36.7 (10.62)

101. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Social Functioning
Description: as for outcome 75
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 36.9 (9.74) | 39.9 (10.07) | 38.3 (10.04) | 38.9 (9.71)

102. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Social Functioning
Description: as for outcome 75
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 37.1 (10.41) | 40.0 (9.60) | 39.0 (10.09) | 40.2 (9.44)

103. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Social Functioning
Description: as for outcome 75
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 37.3 (10.93) | 38.9 (10.01) | 40.2 (10.15) | 39.6 (8.67)

104. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Social Functioning
Description: as for outcome 75
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 37.1 (11.97) | 39.0 (10.77) | 37.2 (10.18) | 38.8 (10.70)

105. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Role-Emotional
Description: as for outcome 75
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 29.3 (12.17) | 31.2 (11.66) | 31.1 (9.96) | 32.7 (13.03)

106. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Role-Emotional
Description: as for outcome 75
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 34.8 (10.88) | 36.2 (12.69) | 34.1 (10.32) | 34.6 (10.96)

107. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Role-Emotional
Description: as for outcome 75
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 33.3 (12.19) | 38.3 (11.79) | 34.5 (11.09) | 36.5 (10.91)

108. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Role-Emotional
Description: as for outcome 75
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 33.4 (12.14) | 37.4 (12.38) | 35.0 (11.46) | 36.5 (11.17)

109. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Role-Emotional
Description: as for outcome 75
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 34.4 (13.11) | 36.4 (10.77) | 35.2 (10.73) | 36.1 (12.46)

110. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Mental Health
Description: as for outcome 75
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 35.3 (12.54) | 37.4 (10.99) | 36.1 (11.39) | 38.9 (12.06)

111. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Mental Health
Description: as for outcome 75
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 40.6 (11.13) | 43.3 (12.95) | 38.9 (12.64) | 40.9 (10.80)

112. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Mental Health
Description: as for outcome 75
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 40.5 (11.70) | 42.9 (12.44) | 39.7 (12.63) | 42.7 (11.43)

113. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Mental Health
Description: as for outcome 75
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 41.0 (11.23) | 43.1 (11.58) | 39.7 (12.14) | 41.7 (11.66)

114. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Mental Health
Description: as for outcome 75
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 40.5 (12.27) | 41.4 (13.00) | 37.7 (11.70) | 40.4 (12.11)

115. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Mental Health Component Score
Description: SF-36V2 is a generic 36-item generic health status measure covering 2 summary measures: physical component summary (PCS) and mental health component score (MCS); it consists of 8 subscales. The MCS is represented by 4 subscales: vitality, social function, role limitations due to emotional problems, and mental health. Participants self-report on items in a subscale that have choices per item. Scoring is done for both MCS subscale scores and summary scores; for each, the range is 0 (worst) to 100 (best).
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 35.9 (12.47) | 37.8 (10.91) | 37.3 (10.11) | 40.0 (11.86)

116. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Mental Health Component Score
Description: The SF-36v2 (Acute version) is a 36-item generic health status measure that yields an 8-scale profile of functional health and well-being as well as psychometrically-based physical and mental health summary measures. The SF-36v2 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. The lower the score the more disability, while the higher the score the less disability. Additionally, two summary scale scores can be calculated: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Summary statistics were calculated for each of the 8 scales, the 2 summary measures, and changes from baseline for each treatment group.
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 41.1 (11.01) | 43.3 (12.95) | 39.9 (11.52) | 40.4 (10.79)

117. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Mental Health Component Score
Description: as for outcome 116
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 40.2 (11.36) | 43.7 (11.41) | 40.6 (12.35) | 42.8 (10.82)

118. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Mental Health Component Score
Description: as for outcome 116
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 40.7 (11.06) | 43.1 (11.31) | 40.9 (11.66) | 41.7 (11.35)

119. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Mental Health Component Score
Description: as for outcome 116
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 40.4 (11.98) | 42.3 (12.10) | 39.3 (11.14) | 41.1 (11.92)

120. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Physical Component Score
Description: as for outcome 116
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 32.1 (6.06) | 32.8 (5.91) | 32.9 (6.30) | 33.9 (6.98)

121. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Physical Component Score
Description: as for outcome 116
Time Frame: Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 35.3 (7.47) | 36.6 (7.73) | 37.1 (7.08) | 40.5 (7.57)

122. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Physical Component Score
Description: as for outcome 116
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 35.8 (7.59) | 38.1 (8.12) | 37.2 (6.73) | 40.0 (8.78)

123. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Physical Component Score
Description: as for outcome 116
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 36.5 (8.26) | 38.3 (8.82) | 38.2 (8.65) | 40.3 (8.16)

124. Secondary Outcome: SF-36 Health Questionnaire - Version 2 (SF-36v2) - Physical Component Score
Description: as for outcome 116
Time Frame: Week 16 (Follow-up)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Number analyzed (Participants) | 49 | 48 | 49 | 50
units on a scale | 37.1 (9.50) | 37.6 (7.34) | 37.2 (7.95) | 39.0 (7.96)

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events (TEAEs) were collected for approximately 1 year. They were collected throughout the duration of the study, which began in April, 2008 and concluded in July, 2009. All patients who were enrolled in the study and received at least one dose of study drug were included in AE reporting.
Description: An AE is any untoward medical occurrence including the exacerbation of a pre-existing condition, in a patient or clinical investigation subject administered a pharmaceutical product. This does not necessarily have a causal relationship with this treatment.
Arm/Group | Placebo | ARRY-438162: 10 mg Bid | ARRY-438162: 40 mg qd | ARRY-438162: 20 mg Bid
Serious Adverse Events (participants affected / at risk) | 1/49 | 1/49 | 1/50 | 0/50
Other Adverse Events (participants affected / at risk) | 20/49 | 25/49 | 39/50 | 42/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | ARRY-438162: 10 mg Bid (N=49) | ARRY-438162: 40 mg qd (N=50) | ARRY-438162: 20 mg Bid (N=50)
BRONCHOPNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEST INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | ARRY-438162: 10 mg Bid (N=49) | ARRY-438162: 40 mg qd (N=50) | ARRY-438162: 20 mg Bid (N=50)
DIARRHOEA (Gastrointestinal disorders) | 5 (5) | 3 (3) | 15 (15) | 12 (12)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANAL FISSURE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEILITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TONGUE DISORDER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HIATUS HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 7 (7) | 5 (5)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
ROSACEA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIVEDO RETICULARIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIORBITAL OEDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PIGMENTATION DISORDER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PLANTAR ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRURIGO (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 4 (4) | 4 (4) | 2 (2) | 5 (5)
BRONCHITIS (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 4 (4)
FOLLICULITIS (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
ACUTE TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GENITAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HELICOBACTER GASTRITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PHARYNGOTONSILLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TRACHEITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TRACHEOBRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASYMPTOMATIC BACTERIURIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 4 (4) | 5 (5) | 5 (5)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
TRANSAMINASES INCREASED (Investigations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
BLOOD PRESSURE SYSTOLIC ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ELECTROCARDIOGRAM REPOLARISATION ABNORMALITY (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 5 (5) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
FACE OEDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
GENERALISED OEDEMA (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
THIRST (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOTONIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VASCULITIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LEFT VENTRICULAR HYPERTROPHY (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EYE SWELLING (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SCOTOMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALLERGIC SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
ABDOMINAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
EXCORIATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
JOINT INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY BLADDER POLYP (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GENITAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SPONTANEOUS HAEMATOMA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of the sponsor's agreements with its investigators may vary. However, the sponsor does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e. data from all sites) in the clinical trial.